CLINICAL TRIAL: NCT06531434
Title: A Pilot Study to Establish Best Treatment Strategy for T4 Esophageal Cancer
Brief Title: Establishing Best Treatment Strategy for T4 Esophageal Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-BR-113-045
Record Dates: First submitted 2024-07-16; First posted 2024-08-01 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-07

CONDITIONS: Esophageal Cancer TNM Staging Primary Tumor (T) T4
Keywords: T4 esophageal cancer; Induction chemotherapy
MeSH Terms: interventions — Docetaxel; Cisplatin; Fluorouracil; Radiation

STUDY DESIGN:
Intervention Model Description: All participants will receive an induction chemotherapy regimen consisting of 4-8 cycles of docetaxel, cisplatin, and fluorouracil. It is followed by concurrent chemoradiotherapy if down-stage had been achieved by induction chemotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Induction chemotherapy followed by chemoradiotherapy (Experimental): This is a single-arm study. All patients will be assigned to receive Induction chemotherapy followed by concurrent chemoradiotherapy.
  Interventions: Combination Product: "Docetaxel", "Cisplatin", "fluorouracil", "Radiation"

INTERVENTIONS:
Combination Product: "Docetaxel", "Cisplatin", "fluorouracil", "Radiation" — Induction chemotherapy with Docetaxel, Cisplatin, and fluorouracil for 4 to 8 cycles, followed by concurrent chemoradiotherapy with Cisplatin and Radiation 30.6-40 Gy.

SUMMARY:
The goal of this clinical trial is to investigate the safety and efficacy of a new treatment approach for T4-stage esophageal cancer, which involves chemoradiotherapy after induction chemotherapy. The main questions it aims to answer are:

* Does the new induction chemotherapy followed by chemoradiation reduce esophageal perforation rate?
* Does the new induction chemotherapy followed by chemoradiation increase treatment response rate and patient survival? Researchers will analyze the above data to see if the new treatment approach works to treat T4 esophageal cancer.

Participants will:

* Receive induction chemotherapy for 4 to 8 cycles, followed by chemoradiation therapy if downstage to T3
* Visit the clinic once every week for checkups and tests
* Keep a diary of their symptoms

DETAILED DESCRIPTION:
The treatment of T4-stage esophageal cancer is challenging because of a high esophageal perforation rate (19%) after concurrent chemoradiotherapy. This research aims to investigate whether a novel sequential chemoradiotherapy approach can improve the treatment response rate and reduce the incidence of esophageal perforation in participants with T4-stage esophageal cancer. The proposed novel treatment strategy involves induction chemotherapy for 4 to 8 cycles. It is followed by concurrent chemoradiotherapy if down-stage had been achieved by induction chemotherapy. The study will be conducted in two phases, starting with a phase I study to determine safety, followed by a phase II study to evaluate overall efficacy. Expected outcomes include improved treatment response rates and reduced esophageal perforation rates in T4-stage esophageal cancer, offering a better treatment option for these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed esophageal squamous cell carcinoma
2. Tumor or lymph nodes invade adjacent organs (T4 stage)
3. Aged between 18-70 years old
4. Patient health status score Eastern Cooperative Oncology Group (ECOG) performance status (PS) <2
5. Hemoglobin ≥ 10 g/L, absolute neutrophil count ≥ 2×10^3/L, platelet count ≥ 100×10^9/L, total bilirubin ≤ 1.5 mg/L, serum transaminases ≤ 105 U/L, creatinine clearance ≥ 40 mL/min.

Exclusion Criteria:

1. Previous chemotherapy history
2. Myocardial infarction within the last three months
3. History of unstable angina, interstitial pneumonia, fibrotic lung disease, or severe emphysema
4. Has other malignancies currently
5. Uncontrolled infection
6. Pregnancy or lactation
7. Perforated esophagus at the time of diagnosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate of the treatment | At week 8, week 16, and 4 weeks after completion of concurrent chemoradiotherapy (CCRT).
  Overall response rate = complete response (CR) rate + partial response (PR) rate.
Duration of response (DOR) | At week 8, week 16, and 4 weeks after completion of CCRT. Thereafter, every 3 months.
  Defined as the time from CR or PR to the time of disease progression or death.

SECONDARY OUTCOMES:
Esophageal perforation rate | At week 8, week 16, and 4 weeks after completion of CCRT. And at anytime when participants suffer from symptoms in suspicious of esophageal perforation, eg. chest pain, hemoptysis, and fever.
  Detected by bronchoscopy or CT scan.
Adverse events of treatment | During treatment (up to 24 weeks)
  Any adverse events of chemotherapy or CCRT.
Progression-free survival | At week 8, week 16, and 4 weeks after completion of CCRT. Thereafter, every 3 months.
  Defined as the time from diagnosis to the time of disease progression or death.
Overall survival time | At week 8, week 16, and 4 weeks after completion of CCRT. Thereafter, every 3 months.
  Defined as the time from diagnosis to the time of death.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared. Results will be published by the investigators in academic journals.

REFERENCES:
- [Background] Chan WL, Choi CW, Wong IY, Tsang TH, Lam AT, Tse RP, Chan KK, Wong C, Law BT, Cheung EE, Chan SY, Lam KO, Kwong D, Law S. Docetaxel, Cisplatin, and 5-FU Triplet Therapy as Conversion Therapy for Locoregionally Advanced Unresectable Esophageal Squamous Cell Carcinoma. Ann Surg Oncol. 2023 Feb;30(2):861-870. doi: 10.1245/s10434-022-12694-8. Epub 2022 Oct 28. PMID 36307666
- [Background] Specht G. [Current problems of surgical diagnosis and surgical treatment of bronchial carcinoma]. Internist (Berl). 1970 Sep;11(9):331-4. No abstract available. German. PMID 4921115
- [Background] Makino T, Yamasaki M, Miyazaki Y, Wada N, Takahashi T, Kurokawa Y, Nakajima K, Takiguchi S, Mori M, Doki Y. Utility of initial induction chemotherapy with 5-fluorouracil, cisplatin, and docetaxel (DCF) for T4 esophageal cancer: a propensity score-matched analysis. Dis Esophagus. 2018 Apr 1;31(4). doi: 10.1093/dote/dox130. PMID 29190316